CLINICAL TRIAL: NCT06360744
Title: A Phase IV Vaccine Study Under the National Cohort Study of Effectiveness and Safety of SARS-CoV-2 (COVID-19) Vaccines (ENFORCE PLUS)
Brief Title: A Phase IV Vaccine Study Under the National Cohort Study of Effectiveness and Safety of SARS-CoV-2 (COVID-19) Vaccines.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jens D Lundgren, MD (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government)
Responsible Party: Sponsor-Investigator, Jens D Lundgren, MD, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ENFORCE PLUS
Record Dates: First submitted 2021-07-01; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: SARS CoV 2 Infection
Keywords: COVID-19; Vaccination
MeSH Terms: conditions — COVID-19 | interventions — Ad26COVS1

STUDY DESIGN:
Intervention Model Description: The design is an open-labelled, non-randomised, parallel group, phase IV study with historical controls.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccine Johnson and Johnson/Janssen Covid-19 vaccine (Other): Johnson & Johnson/Janssen Covid-19 vaccine.
  Interventions: Biological: Johnson & Johnson

INTERVENTIONS:
Biological: Johnson & Johnson — Vaccination with the Johnson & Johnson vaccine which is NOT part of the Danish National Government programme

SUMMARY:
A phase IV study to assess if the SARS-CoV-2 vaccine from Johnson & Johnson/Janssen (J&J) results in change in number and activation of platelets and anti-PF4 Level. As well as compare whether the vaccine is causing a greater activation of platelets and anti-PF4 than the mRNA vaccines.

The Danish Medicines Agency has approved the vaccine from J&J for use in Denmark, however it is not currently part of the national vaccine programme.

The design is an open-labelled, non-randomised, parallel group, phase IV study with historical controls. A sub-study will be embedded within this master protocol addressing basic and translational research questions requiring additional sampling of biological material (under separate participant informed consent).

DETAILED DESCRIPTION:
Participants will have 3 specific study visits and will hereafter be followed for 2 years after the vaccination with regular visits after 3, 6, 12 and 24 month. In this way the participants will be offered an extra close follow up on vaccine effectiveness.

Safety data will be collected at study visits until 3 months after the first vaccination,, with additional safety data collected under this protocol during the first month after vaccination.

Research samples will be collected at each study visit during the two-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before any trial related procedures are performed
2. Male or female eligible for SARS-CoV-2 immunization (as defined by SST in the 'Tilvalgsordningen')
3. The subject must be willing and able to comply with trial protocol (re-visits and biological samples)

Exclusion Criteria:

1. Male and female under the age of 18
2. Any subgroup of individuals for which the vaccine is contra-indicated
3. Previous SARS-CoV-2 vaccination

   Specific for the Johnson & Johnson vaccine:
4. Experience of a serious allergic reaction after injection of any other vaccine
5. Serious infection with high fever (> 38 0C) A temporary postponement of the vaccination is allowed, when participant has been well for at least 48 hours. Mild fever or upper airway infection like a cold is not a problem
6. Problems with bleeding or bruising, or use of anticoagulant medicine (to prevent blood clots)
7. Immunodeficiency or use of medicines that weaken the immune system (such as high-dose corticosteroids, immunosuppressants or cancer medicines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the J& J vaccine | The change from base-line to after 24 month
  To clarify whether vaccination with the J&J vaccine leads to changes in the number and activation of platelets as well as anti-PF4 level and to compare whether the J&J vaccine causes a stronger activation of platelets as well as an increase in anti-PF4 antibodies compared to mRNA vaccines. Included is also questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jens Lundgren, Professor, Study Chair — Rigshospitalet, Denmark
Locations (5):
- Denmark (5):
  - Aarhus Universitetshospital, Skejby, Aarhus, Aarhus N
  - Aalborg Universitetshospital Syd, Aalborg
  - Hvidovre Hospital, Hvidovre
  - Odense Universitetshospital, Odense
  - Sjællandsuniversitetshospital, Roskilde

IPD SHARING:
Plan to Share IPD: No